CLINICAL TRIAL: NCT03959852
Title: A Combination Study With Sub-Dissociative Ketamine and Fentanyl to Treat Moderate to Severe Pain in the Emergency Department
Brief Title: Sub-Dissociative Ketamine and Fentanyl to Treat Moderate to Severe Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Residency completed.
Sponsor: Mercy Health Ohio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-040
Record Dates: First submitted 2019-03-12; First posted 2019-05-22 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Pain, Acute
Keywords: Moderate; Severe; Pain
MeSH Terms: conditions — Acute Pain; Lymphoma, Follicular; Pain | interventions — Fentanyl; Ketamine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sub-Dissociative Ketamine alone (Active Comparator): 0.3 mg/kg of Sub-Dissociative Ketamine IV administered over at least 1 minute
  Interventions: Drug: Ketamine
- Fentanyl alone (Active Comparator): 1 mg/kg of Fentanyl IV administered over at least 1 minute
  Interventions: Drug: Fentanyl
- Sub-dissociative Ketamine and Fentanyl (Experimental): Combined dose of 0.15 mg/kg of Sub-dissociative Ketamine and 0.5 mg/kg of Fentanyl IV administered over at least 1 minute
  Interventions: Combination Product: Fentanyl and Ketamine

INTERVENTIONS:
Drug: Fentanyl — 1 mg/kg of Fentanyl IV administered over at least 1 minute
  Other Names: Fentanyl Citrate
  Arms: Fentanyl alone
Combination Product: Fentanyl and Ketamine — Combined dose of 0.15 mg/kg of Sub-dissociative Ketamine and 0.5 mg/kg of Fentanyl IV administered over at least 1 minute.
  Arms: Sub-dissociative Ketamine and Fentanyl
Drug: Ketamine — 0.3 mg/kg of Sub-Dissociative Ketamine IV administered over at least 1 minute
  Other Names: Ketamine Hydrochloride
  Arms: Sub-Dissociative Ketamine alone

SUMMARY:
The objective of this study is to evaluate the potential opioid-sparing effect associated with the novel combination of fentanyl and sub-dissociative ketamine in adult patients with moderate to severe pain in the emergency department.

DETAILED DESCRIPTION:
Pain is a very common complaint in the emergency department (ED). The use of opioids to treat moderate to severe pain has increased over the last decade as well as the number of opioid related deaths. In 1999 to 2016, more than 630,000 people died from a drug overdose. Treatment for acute pain has been assessed in the ED, with review of several different pain medications. Sub-dissociative ketamine (SDK) has become a valuable treatment option for acute pain and in recent years, has been of increased interest due to the growing concerns regarding opioid abuse and opioid shortage in the United States. Sub-dissociative ketamine, an NMDA receptor antagonist, has been studied in dose ranges of 1-4.5 mg/kg for dissociative sedation, as well as dose ranges of 0.1-0.3 mg/kg to treat pain. The onset of action for an IV dose of 2 mg/kg has been studied, with onset usually within 30 seconds after injection and anesthetic effect lasting 5-10 minutes. Common side effects include elevated blood pressure, diplopia or nystagmus, nausea and vomiting. More rare and more severe side effects in dissociative doses include respiratory depression, emergency phenomenon, tonic and clonic movements, and anaphylaxis. However, these were rarely, if ever seen, findings in sub-dissociative doses. Several studies indicate that SDK is a safe and effective alternative to opioids for patients with complaints of moderate to severe pain that provides adequate analgesic effect by itself. In particular, several studies have compared SDK versus morphine, particularly looking at pain in individuals with abdominal pain, flank pain, low back pain or musculoskeletal pain, and acute fractures. SDK has also shown to decrease opioid consumption and the need for rescue analgesia. The studies showed that that there was no difference in average pain scores, but the amount of morphine required was significantly decreased. SDK has proven to be a safe alternative, but the side effects, although short, make it less desirable to use. To the investigator's knowledge, there has never been a study focusing on the use of combination fentanyl and SDK. Fentanyl, an opioid agonist, has been studied in low dose forms of 2 mcg/kg for pain, moderate dose forms of 2-20 mcg/kg for major surgical procedures, and high dose forms of 20-50 mcg/kg for orthopedic and open heart surgeries. Onset of action is almost immediate when given IV, and maximal effect of the drug may take several minutes. The usual duration of action is 30-60 minutes. Common side effects include hypertension, hypotension, dizziness, blurred vision, nausea, vomiting and laryngospasm. Serious side effects included respiratory depression, apnea, rigidity, bradycardia, serotonin syndrome, adrenal insufficiency, and if left untreated could cause cardiac arrest and circulatory depression. There have been several combination studies with SDK, but none regarding fentanyl and ketamine. In one study, combination SDK and reduced dose hydromorphone produced rapid pain relief without significant side effects. Another study indicated that morphine and SDK both provided adequate pain relief alone, but combined morphine and SDK required less morphine administration, had faster onset of relief, and provided sustained reduction in pain intensity for up to 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years old
* Moderate pain defined as 4-6 out of 10, severe pain defined as ≥ 7 out of 10 as defined by the numeric rating pain scale (NRS)
* Proficient in reading and understanding English
* Are deemed by the attending physician to require opioid therapy.

Exclusion Criteria:

* Inability to give consent,
* Inability to use the numeric rating scale (NRS) score
* Long-term use of opioids, history of chronic pain
* Known substance abuse known as excessive use of a drug such as (e.g. alcohol, narcotics or cocaine)
* Known hypersensitivity to ketamine or fentanyl
* Pregnancy
* Alcohol intoxication
* Depression
* Anxiety
* Chronic obstructive pulmonary disease
* Asthma
* Cirrhosis
* On dialysis
* Acute ischemic stroke
* Heart rate (HR) less < 60 bpm or > 120 bpm
* Systolic blood pressure (SBP) < 90 mmHg or > 180 mmHg
* Ischemic heart disease
* Ketamine prior to arrival
* Trauma patients
* Sepsis or septic shock
* Weight > 100 kg.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
Analgesia of combination fentanyl and SDK as assessed using the pain scale 1-10 | ED encounter (less than 24 hours)
  Analgesia of combination fentanyl and SDK as assessed using the pain scale 1-10
Analgesia of fentanyl as assessed using the pain scale 1-10 | ED encounter (less than 24 hours)
  Analgesia of fentanyl as assessed using the pain scale 1-10
Analgesia of ketamine as assessed using the pain scale 1-10 | ED encounter (less than 24 hours)
  Analgesia of katamine as assessed using the pain scale 1-10

SECONDARY OUTCOMES:
OARRS report | ED encounter (less than 24 hours)
  A retrospective review of OARRS report will be performed with each patient.
Opioid sparing response as assessed by number of times additional rescue doses of fentanyl were required | ED encounter (less than 24 hours)
  Opioid sparing response as assessed by number of times additional rescue doses of fentanyl were required

CONTACTS AND LOCATIONS:
Overall Officials: David Gemmel, Study Director — Director of Research
Locations (1):
- St. Elizabeth Boardman Hospital, Boardman, Ohio, United States

REFERENCES:
- [Background] Hebsgaard S, Mannering A, Zwisler ST. Assessment of acute pain in trauma-A retrospective prehospital evaluation. J Opioid Manag. 2016 Sep/Oct;12(5):347-353. doi: 10.5055/jom.2016.0351. PMID 27844474
- [Background] Motov SM, Nelson LS. Advanced Concepts and Controversies in Emergency Department Pain Management. Anesthesiol Clin. 2016 Jun;34(2):271-85. doi: 10.1016/j.anclin.2016.01.006. PMID 27208710
- [Background] Todd KH. A Review of Current and Emerging Approaches to Pain Management in the Emergency Department. Pain Ther. 2017 Dec;6(2):193-202. doi: 10.1007/s40122-017-0090-5. Epub 2017 Nov 10. PMID 29127600
- [Background] Bowers KJ, McAllister KB, Ray M, Heitz C. Ketamine as an Adjunct to Opioids for Acute Pain in the Emergency Department: A Randomized Controlled Trial. Acad Emerg Med. 2017 Jun;24(6):676-685. doi: 10.1111/acem.13172. Epub 2017 Mar 22. PMID 28177167
- [Background] Duncan C, Riley B. BET 2: Low-dose ketamine for acute pain in the ED. Emerg Med J. 2016 Dec;33(12):892-893. doi: 10.1136/emermed-2016-206440.2. PMID 27864394
- [Background] Jennings PA, Cameron P, Bernard S, Walker T, Jolley D, Fitzgerald M, Masci K. Long-term pain prevalence and health-related quality of life outcomes for patients enrolled in a ketamine versus morphine for prehospital traumatic pain randomised controlled trial. Emerg Med J. 2014 Oct;31(10):840-3. doi: 10.1136/emermed-2013-202862. Epub 2013 Jul 13. PMID 23851034
- [Background] Lee EN, Lee JH. The Effects of Low-Dose Ketamine on Acute Pain in an Emergency Setting: A Systematic Review and Meta-Analysis. PLoS One. 2016 Oct 27;11(10):e0165461. doi: 10.1371/journal.pone.0165461. eCollection 2016. PMID 27788221
- [Background] Miller JP, Schauer SG, Ganem VJ, Bebarta VS. Low-dose ketamine vs morphine for acute pain in the ED: a randomized controlled trial. Am J Emerg Med. 2015 Mar;33(3):402-8. doi: 10.1016/j.ajem.2014.12.058. Epub 2015 Jan 7. PMID 25624076
- [Background] Motov S, Rockoff B, Cohen V, Pushkar I, Likourezos A, McKay C, Soleyman-Zomalan E, Homel P, Terentiev V, Fromm C. Intravenous Subdissociative-Dose Ketamine Versus Morphine for Analgesia in the Emergency Department: A Randomized Controlled Trial. Ann Emerg Med. 2015 Sep;66(3):222-229.e1. doi: 10.1016/j.annemergmed.2015.03.004. Epub 2015 Mar 26. PMID 25817884
- [Background] Motov S, Rosenbaum S, Vilke GM, Nakajima Y. Is There a Role for Intravenous Subdissociative-Dose Ketamine Administered as an Adjunct to Opioids or as a Single Agent for Acute Pain Management in the Emergency Department? J Emerg Med. 2016 Dec;51(6):752-757. doi: 10.1016/j.jemermed.2016.07.087. Epub 2016 Sep 29. PMID 27693070
- [Background] Pourmand A, Mazer-Amirshahi M, Royall C, Alhawas R, Shesser R. Low dose ketamine use in the emergency department, a new direction in pain management. Am J Emerg Med. 2017 Jun;35(6):918-921. doi: 10.1016/j.ajem.2017.03.005. Epub 2017 Mar 2. PMID 28285863
- [Background] Sin B, Ternas T, Motov SM. The use of subdissociative-dose ketamine for acute pain in the emergency department. Acad Emerg Med. 2015 Mar;22(3):251-7. doi: 10.1111/acem.12604. Epub 2015 Feb 25. PMID 25716117
- [Background] Abbasi S, Bidi N, Mahshidfar B, Hafezimoghadam P, Rezai M, Mofidi M, Farsi D. Can low-dose of ketamine reduce the need for morphine in renal colic? A double-blind randomized clinical trial. Am J Emerg Med. 2018 Mar;36(3):376-379. doi: 10.1016/j.ajem.2017.08.026. Epub 2017 Aug 14. PMID 28821365
- [Background] Ahern TL, Herring AA, Miller S, Frazee BW. Low-Dose Ketamine Infusion for Emergency Department Patients with Severe Pain. Pain Med. 2015 Jul;16(7):1402-9. doi: 10.1111/pme.12705. Epub 2015 Feb 3. PMID 25643741
- [Background] Dickenson AH. NMDA receptor antagonists: interactions with opioids. Acta Anaesthesiol Scand. 1997 Jan;41(1 Pt 2):112-5. doi: 10.1111/j.1399-6576.1997.tb04624.x. PMID 9061093
- [Background] Galinski M, Dolveck F, Combes X, Limoges V, Smail N, Pommier V, Templier F, Catineau J, Lapostolle F, Adnet F. Management of severe acute pain in emergency settings: ketamine reduces morphine consumption. Am J Emerg Med. 2007 May;25(4):385-90. doi: 10.1016/j.ajem.2006.11.016. PMID 17499654
- [Background] Lilius TO, Jokinen V, Neuvonen MS, Niemi M, Kalso EA, Rauhala PV. Ketamine coadministration attenuates morphine tolerance and leads to increased brain concentrations of both drugs in the rat. Br J Pharmacol. 2015 Jun;172(11):2799-813. doi: 10.1111/bph.12974. PMID 25297798
- [Background] Wiesenfeld-Hallin Z. Combined opioid-NMDA antagonist therapies. What advantages do they offer for the control of pain syndromes? Drugs. 1998 Jan;55(1):1-4. doi: 10.2165/00003495-199855010-00001. PMID 9463786
- [Background] Ahern TL, Herring AA, Stone MB, Frazee BW. Effective analgesia with low-dose ketamine and reduced dose hydromorphone in ED patients with severe pain. Am J Emerg Med. 2013 May;31(5):847-51. doi: 10.1016/j.ajem.2013.02.008. Epub 2013 Apr 18. PMID 23602757
- [Background] Ahmadi O, Isfahani MN, Feizi A. Comparing low-dose intravenous ketamine-midazolam with intravenous morphine with respect to pain control in patients with closed limb fracture. J Res Med Sci. 2014 Jun;19(6):502-8. PMID 25197290
- [Background] Beaudoin FL, Lin C, Guan W, Merchant RC. Low-dose ketamine improves pain relief in patients receiving intravenous opioids for acute pain in the emergency department: results of a randomized, double-blind, clinical trial. Acad Emerg Med. 2014 Nov;21(11):1193-202. doi: 10.1111/acem.12510. PMID 25377395
- [Background] Bossard AE, Guirimand F, Fletcher D, Gaude-Joindreau V, Chauvin M, Bouhassira D. Interaction of a combination of morphine and ketamine on the nociceptive flexion reflex in human volunteers. Pain. 2002 Jul;98(1-2):47-57. doi: 10.1016/s0304-3959(01)00472-9. PMID 12098616
- [Background] Jennings PA, Cameron P, Bernard S, Walker T, Jolley D, Fitzgerald M, Masci K. Morphine and ketamine is superior to morphine alone for out-of-hospital trauma analgesia: a randomized controlled trial. Ann Emerg Med. 2012 Jun;59(6):497-503. doi: 10.1016/j.annemergmed.2011.11.012. Epub 2012 Jan 13. PMID 22243959
- [Background] Johansson P, Kongstad P, Johansson A. The effect of combined treatment with morphine sulphate and low-dose ketamine in a prehospital setting. Scand J Trauma Resusc Emerg Med. 2009 Nov 27;17:61. doi: 10.1186/1757-7241-17-61. PMID 19943920
- See also: U.S. Department of Health and Human Services. (2018, October 15). U.S. Food and Drug Administration. Retrieved October 15, 2018, from https://www.accessdata.fda.gov/scripts/drugshortages/ — https://www.accessdata.fda.gov/scripts/drugshortages/